CLINICAL TRIAL: NCT01740726
Title: Randomized Trial of Behavioral Activation and Antidepressant Medication in the Treatment of Adolescents With Major Depression
Brief Title: Comparison of Behavioral Activation and Antidepressant Medication in the Treatment of Adolescents With Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of success with recruitment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, W. Edward Craighead, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00061525; CAMP-61525 (Other: Other)
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2015-03

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Behavioral Activation; Fluoxetine; Prozac; Treatment; Therapy; Psychotherapy; Antidepressant; Intervention
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Activation (Experimental)
  Interventions: Behavioral: Behavioral Activation
- Fluoxetine (Active Comparator)
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Behavioral: Behavioral Activation — 18 weeks of 1-hour individual therapy focused on increasing rewarding behaviors. Therapy follows Behavioral Activation manual supported through previous research of this therapy for adolescents. BA intervention includes monthly booster sessions offered throughout 6-month follow up.
  Other Names: Behavioral Activation Therapy; BA
  Arms: Behavioral Activation
Drug: Fluoxetine — Initial 10mg dose titrated as necessary to 40mg daily; weekly visits for 4 weeks, biweekly visits for next 6 weeks, monthly visits for remaining 8 weeks of active treatment and through 6-month follow up. Therapists will be available between sessions and throughout the follow-up interval to manage clinical concerns or emergencies.
  Other Names: Prozac; Sarafem; Rapiflux; Selfemra
  Arms: Fluoxetine

SUMMARY:
This study focuses on treating adolescents with depression. The study has two main purposes. The first is to compare a new form of therapy for depression called Behavioral Activation (BA) to the antidepressant medication fluoxetine. BA therapy helps depressed people get more involved in activities they find enjoyable, which can reduce symptoms of depression. Research shows that both BA and fluoxetine work to reduce depressive symptoms in adolescents. However, unlike previous research, this study examines how well the two treatment options work in comparison to each other. Participants in the study are randomized to receive treatment with either BA or fluoxetine for 18 weeks.

The second aim of the study is to examine the brain functions of adolescents in both treatment groups. Participants undergo functional Magnetic Resonance Imaging (fMRI) scans before and after treatment. The data from these scans will be used to compare the brains of participants in the BA condition with those in the fluoxetine condition. Also, the scans may show possible differences between participants' brains before and after treatment. These data may help scientists determine the ideal form of depression treatment for different types of people.

DETAILED DESCRIPTION:
Depression is a serious diagnosis that can have severe consequences; it is not just experiencing "the blues" or having sad feelings that most people get from time to time. People who are diagnosed with depression have overwhelming feelings of sadness that are present for at least two weeks. In addition, they also experience symptoms such as changes in their appetite or sleep patterns, feelings of guilt or worthlessness, lack of energy or motivation, and even thoughts of suicide. People with depression have difficulty functioning in many areas of their lives, including at work, at school, and in social relationships. Those who have this diagnosis often need medication, therapy, or a combination of both to relieve their symptoms and regain their usual functioning.

This study investigates whether a type of psychotherapy called Behavioral Activation (BA) is as effective as antidepressant medication in the treatment of adolescents diagnosed with depression. In this study, BA is compared to fluoxetine, which is known to help treat depressive symptoms in this population. BA has been shown to be efficacious in reducing depression in adolescents, but it is not yet known how it compares to another leading treatment for depression in this age group. Thus, this study's primary goal is to see how BA compares to fluoxetine.

This study also examines brain activity as it relates to depression and treatment. The study includes functional Magnetic Resonance Imaging (fMRI) scans of participants in both conditions before and after they undergo treatment. Participants play a game in the scanner called the Monetary Incentive Delay (MID) task, and they have the opportunity to win money (reward) or to avoid losing money (loss). After they play the MID game, the scan images show certain brain regions that are activated in reward and loss situations. This study looks at how these brain regions relate to treatment response, especially because the goal of BA is to help people enjoy rewards more. The study also compares brain activity between the two treatment groups, as well as changes in brain activity from pre- to post-treatment. This part of the study should provide information about which kinds of people respond to which kinds of treatment.

Behavioral activation is a new therapy that has been shown to successfully treat depressed adults and adolescents. BA is a type of therapy that helps depressed people get involved in activities that they find to be enjoying and rewarding. The developers of this therapy believe that people are depressed because they are not experiencing rewarding and positive events in their lives very often. For example, when people become depressed, they usually become isolated from others. They also stop doing the things they used to enjoy, or they do them far less often. As a result, they have fewer experiences that make them feel a sense of accomplishment and happiness, and their depression becomes more severe. The worse the symptoms get, the less they engage in rewarding activities. The developers of BA have established a therapy program that helps the patient choose and participate in activities that are rewarding. The therapist acts as a coach, monitoring progress and giving feedback about these activities and the relationship between this activation and mood. This type of therapy is not just designed to get depressed people to do more; rather, time is spent choosing and evaluating specific activities that are particularly rewarding for the client and evaluating the outcome of these activities. Although BA is a novel intervention, early evidence shows that BA is effective with regard to alleviating symptoms of depression. In addition, the results of these studies show that it works in a relatively short amount of time (approximately four months).

Because so little is known about effective psychosocial treatments for depressed adolescents, and because of the risks associated with treating adolescents with medications, it is important to work on developing and supporting new treatments for this at-risk population. The aim of this pilot study is to generate knowledge for both the scientific community and for clinicians by gaining new insight into what works for depressed teens. To accomplish these goals, this study will treat 20 adolescents who meet criteria for Major Depressive Disorder with 18 weeks of therapy or medication. Ten adolescents will be assigned to the BA condition, and 10 will be assigned to the fluoxetine condition. Those in the medication condition will visit with their psychiatrist regularly but will not receive psychotherapy. Those who receive BA will receive between 18 and 20 sessions of therapy.

It is important to note that people are experiencing first episodes of depression at younger and younger ages; hence, rates of depression are rising in younger age groups. Also, suicide is the third leading cause of death among adolescents, and depression is associated with increased thoughts of suicide and suicide attempts. Depressed children and adolescents are more likely to develop a host of other problems, such as substance abuse, and they are more likely to report experiencing stressful life events. For all these reasons, it is important that scientists work to develop therapies that relieve depression in this population. Studies such as this one can help advance knowledge about how best to treat this dangerous illness.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents ages 13-17
* Current diagnosis of Major Depressive Disorder as determined by the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS-PL), Children's Depression Rating Scale (CDRS-R) raw score > 45 (T-score > 65) at baseline
* Estimated full scale IQ > 80 as determined by the Wechsler Intelligence Scale for Children (WISC)
* Able to receive outpatient care
* Willing to discontinue other psychosocial treatments
* Not taking psychotropic medications in the one month prior to consent, with the exception of psychostimulant medication prescribed for the treatment of attention-deficit/hyperactivity disorder (ADHD)

Exclusion Criteria:

* Current or past diagnosis of bipolar, schizophrenia, schizophreniform, schizoaffective disorders, or psychosis not otherwise specified
* Current diagnosis of developmental disorder, severe conduct disorder, life-threatening anorexia, obsessive-compulsive disorder, or autism-spectrum disorders
* Taking psychotropic medications prior to entry
* Estimated IQ < 80
* Alcohol/drug dependence or abuse within the last 3 months
* Potential/confirmed neurological disorder or epilepsy
* Claustrophobia
* Presence of a medical condition that precludes fMRI
* Endorsement of imminent and serious suicidality
* Medical conditions for which treatment with fluoxetine is contraindicated or that take precedence over the presence of major depressive disorder (MDD)
* Pregnancy

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Craighead, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Executive Park, Atlanta, Georgia, United States

REFERENCES:
- [Background] Ritschel, L. A., Ramirez, C. L., Jones, M., & Craighead, W. (2011). Behavioral activation for depressed teens: A pilot study. Cognitive And Behavioral Practice, 18(2), 281-299. doi:10.1016/j.cbpra.2010.07.002
- [Background] Jacob M, Keeley ML, Ritschel L, Craighead WE. Behavioural activation for the treatment of low-income, African American adolescents with major depressive disorder: a case series. Clin Psychol Psychother. 2013 Jan-Feb;20(1):87-96. doi: 10.1002/cpp.774. Epub 2011 Aug 22. PMID 21861272
- See also: Related Info — http://www.camp-emory.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were screen failures and were not randomized into either arm of the study.
Period: Overall Study
Arm/Group | Behavioral Activation | Fluoxetine
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis is only for the subject that completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation | Fluoxetine | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 1 | 1
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms From Baseline Based on Beck Depression Inventory, 2nd Edition (BDI-II)
Description: Self-report measure, completed by the child, that assesses depressive symptom severity. The BDI-II total score ranges from 0 to 63, with a higher score indicating a higher level of depression. Change is the difference between the 42 week score and the baseline score.
Time Frame: Baseline, 42 weeks
Measure: Number; unit: units on a scale
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 1
units on a scale |  | -45

2. Primary Outcome: Change in Depressive Symptoms From Baseline Based on Children's Depression Rating Scale - Revised (CDRS-R)
Description: Interview-based measure, completed with both the parent and child, that assesses depression severity.
Time Frame: Baseline, 9 wks., 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Improvement and Change in Symptom Severity From Baseline Based on Clinical Global Impression - Improvement and Severity (CGI-I, CGI-S)
Description: Clinician's rating of symptom severity and improvement since baseline.
Time Frame: Baseline, 9 wks., 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Behaviors From Baseline Based on Behavioral Activation for Depression Scale (BADS)
Description: Assesses behavioral changes on 4 subscales: Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment.
Time Frame: Baseline, 9 wks., 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Anxiety From Baseline Based on Multidimensional Anxiety Scale for Children (MASC)
Description: Measures anxiety symptom severity.
Time Frame: Baseline, 9 wks., 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Suicidal Ideation Based on Suicidal Ideation Questionnaire (SIQ)
Description: Assesses seriousness of suicidal intent.
Time Frame: Baseline, 9 wks., 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Hope Based on Children's Hope Scale (CHS)
Description: Assesses self-perception of ability to set and work toward goals.
Time Frame: Baseline, 9 wks., 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Adolescent Longitudinal Interval Follow-up Evaluation (A-LIFE)
Description: Semi-structured interview that assesses psychiatric symptoms, treatments, and functional outcomes in the time period that has elapsed since the previous assessment and tracks change over time.
Time Frame: 18 wks., 30 wks, 42 wks
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Child's Behavior Checklist - Parent Version (CBCL-P)
Description: Completed by parents to describe the child's behavioral and emotional difficulties. Scores reflect observed problems and level of adaptive functioning.
Time Frame: 18 wks., 30 wks., 42 wks.
Population: Data are not available for analysis.
Arm/Group | Behavioral Activation | Fluoxetine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Behavioral Activation | Fluoxetine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The study terminated early due to difficulties with enrolling participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No